CLINICAL TRIAL: NCT06272071
Title: A Multicenter Prospective Clinical Cohort Study on the Pathogen Spectrum of Severe Hepatitis (Liver Failure) Complicated With Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Beijing Ditan Hospital (Other); Beijing YouAn Hospital (Other); Huashan Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Jiajia Chen, Chief Physician of the First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang University
Other Study IDs: 2023YFC2308802-01
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Liver Failure
Keywords: Severe hepatitis; Pathogen pedigree of infection; cohort study
MeSH Terms: conditions — Liver Failure; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — According to the characteristics of infection, take blood or body fluids from the corresponding infected site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to expound the population and characteristics of pathogenic microorganisms with co-infection, draw the pedigree of pathogenic microorganisms, and evaluate its influence on disease outcome in patients with severe hepatitis (liver failure). The main questions it aims to answer are:

* Mapping of infectious agents in patients with severe hepatitis (liver failure)
* Constructing early warning predictive models to explore how to give an individualized regimen of integrated immune function.

DETAILED DESCRIPTION:
Liver failure is a clinical syndrome caused by a large number of necrotic hepatocytes leading to severe liver function damage, with jaundice, coagulation dysfunction and hepatic encephalopathy as the main manifestations, which can be caused by a variety of reasons, and the liver failure caused by Hepatitis B Virus (HBV) is the first one in our country, which accounts for about 80% of the cases. Through the "Eleventh Five-Year Plan" to "Thirteenth Five-Year Plan" national scientific and technological major special projects, the death rate of patients with early and middle stage of severe hepatitis B has been significantly reduced, but the death rate of patients with advanced stage is still as high as about 60%, especially when liver failure is combined with other complications, such as This study focuses on the impact of secondary infections on the clinical prognosis of severe hepatitis (liver failure), and intends to establish a prospective, multi-center clinical cohort of secondary infections in liver failure, map the infectious pathogens, correlate the basic immune status with the characteristics of the pathogen profile of the secondary infections, and establish a monitoring and early-warning system of secondary infections, so as to explore safe and effective treatment modalities. To further reduce the mortality rate of liver failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients agreed to participate in the study and signed an informed consent form;
2. Sex is not limited and age is 18-70 years old;
3. HBsAg positive for more than 6 months, or hepatitis E IgM positive, or hepatitis E RNA positive;
4. Progressive deepening of jaundice in a short period of time (serum total bilirubin greater than 10 times the upper limit of normal or rising ≥17.1 umol/L per day);
5. Sgnificant bleeding tendency with PTA ≤ 40% and exclusion of other non-hepatic factors.

Exclusion Criteria:

1. Patients with severe hepatitis caused by other non-hepatophilic viral infections;
2. Patients who were considered by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe viral hepatitis (liver failure) who met the inclusion and exclusion criteria and were hospitalized in the First Hospital Affiliated to Zhejiang University School of Medicine, Beijing Ditan Hospital Affiliated to Capital Medical University, Beijing You'an Hospital Affiliated to Capital Medical University, Huashan Hospital Affiliated to Fudan University, and Qilu Hospital of Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of secondary infections in patients with severe viral hepatitis (liver failure) at 4 weeks, including site of infection and pathogen of infection. | 4 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or Next-generation sequencing(NGS) results.
quick SEPSIS RELATED ORGAN FAILURE ASSESSMENT(qSOFA) at 4 weeks | 4 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.

SECONDARY OUTCOMES:
Occurrence of secondary infections in patients with severe viral hepatitis (liver failure) at 8 weeks, including site of infection and pathogen of infection. | 8 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or NGS results.
Occurrence of secondary infections in patients with severe viral hepatitis (liver failure) at 12 weeks, including site of infection and pathogen of infection. | 12 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or NGS results.
qSOFA score at 8 weeks | 8 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.
qSOFA score at 12 weeks | 12 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.

CONTACTS AND LOCATIONS:
Overall Officials: Jiajia Chen, Principal Investigator — Zhejiang University